CLINICAL TRIAL: NCT02258542
Title: A Multicentre, Double-blind, Randomized, Parallel Group, Phase 3 Safety Extension Study to Evaluate the Safety and Tolerability of Benralizumab (MEDI-563) in Asthmatic Adults and Adolescents on Inhaled Corticosteroid Plus Long-acting β2 Agonist (BORA)
Brief Title: A Safety Extension Study to Evaluate the Safety and Tolerability of Benralizumab (MEDI-563) in Asthmatic Adults and Adolescents on Inhaled Corticosteroid Plus LABA
Acronym: BORA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: D3250C00021; U1111-1162-2422 (Other: WHO)
Record Dates: First submitted 2014-09-01; First posted 2014-10-07 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: Asthma, Bronchial Diseases, Respiratory Tract Diseases, Lung Diseases, Obstructive Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Benralizumab Arm A (Experimental): Benralizumab administered subcutaneously
  Interventions: Biological: Benralizumab
- Benralizumab Arm B (Experimental): Benralizumab administered subcutaneously
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Benralizumab administered subcutaneously
  Arms: Benralizumab Arm A
Biological: Benralizumab — Benralizumab administered subcutaneously
  Arms: Benralizumab Arm B

SUMMARY:
The purpose of this study is to characterize the safety profile of benralizumab administration in asthma patients who have completed one of the three predecessor studies: D3250C00017, D3250C00018 or D3250C00020.

DETAILED DESCRIPTION:
After a minimum of 1200 patients have been enrolled in this study, subsequent patients (up to a maximum of 2200 total for the study), who complete a minimum of 16 weeks, and no more than 40 weeks, in this study, will be given the option to transition to an open-label safety extension study, Study D3250C00037 (MELTEMI).

Adolescent patients, patients from Japan and South Korea, and any patient who chooses not to enter Study D3250C00037 will remain in this study through IPD or EOT and FU.

At the time of the first interim analysis in Japanese patients, the study regimen for all patients will become unblinded to AstraZeneca for data analysis purposes. Study conduct and blinding at the site and patient level will remain unchanged.

ELIGIBILITY:
Inclusion criteria

1. Informed consent (and/or assent as applicable locally) for study participation must be obtained prior to any study related procedures being performed (local regulations are to be followed in determining the assent/consent requirements for children and parent(s)/guardian(s)) and according to international guidelines and/or applicable European Union guidelines.
2. Female and male patients who completed the double-blind treatment period in a predecessor study on benralizumab or matching placebo.
3. Women of childbearing potential (WOCBP) must agree to use an effective form of birth control throughout the study duration and for 16 weeks after last dose of Investigational Product (IP).
4. For WOCBP only: Have a negative urine pregnancy test prior to administration of Investigational Product (IP) at Visit 1.
5. All male patients who are sexually active must agree to use a double barrier method of contraception (condom with spermicide) from the first dose of IP until 16 weeks after their last dose.

Exclusion criteria

1. Any disorder including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric or major physical impairment that is not stable in the opinion of the Investigator and could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the studies or their interpretations
   * Impede the patient's ability to complete the entire duration of study
2. A helminth parasitic infection diagnosed during a predecessor study that has either not been treated, has been incompletely treated or has failed to respond to standard of care therapy
3. Any clinically significant change in physical examination, vital signs, electrocardiogram (ECG), haematology, clinical chemistry, or urinalysis during a predecessor study which in the opinion of the investigator may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or interfere with the patient's ability to complete the entire duration of the study
4. Current malignancy or malignancy that developed during a predecessor study (subjects that had basal cell carcinoma, localized squamous cell carcinoma of the skin which was resected for cure, or in situ carcinoma of the cervix that has been treated/cured will not be excluded).
5. Receipt of live attenuated vaccines within 30 days prior to initiation of treatment in this study, during the treatment period, and for 16 weeks (5 half-lives) after the last dose of the investigational product
6. Receipt of immunoglobulin or blood products within 30 days prior to Visit 1
7. Planned major surgical procedures during the conduct of the study
8. Previous participation in the present study
9. Concurrent enrolment in another clinical trial
10. AstraZeneca staff involved in the planning and/or conduct of the study
11. Employees of the study centre or any other individuals involved with the conduct of the study or immediate family members of such individuals
12. Patients with major protocol deviations in any of the predecessor studies at the discretion of the Sponsor

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2133 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W. Busse, M.D., Professor of Medicine, Principal Investigator — Allergy, Pulmonary, and Critical Care Medicine 600 Highland Avenue; Madison, WI
Locations (328):
- United States (83):
  - Research Site, Andalusia, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsboro, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Alhambra, California
  - Research Site, Bakersfield, California
  - Research Site, Newport Beach, California
  - Research Site, Redondo Beach, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Jose, California
  - Research Site, Stockton, California
  - Research Site, Walnut Creek, California
  - Research Site, Westminster, California
  - Research Site, Woodland, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Cutler Bay, Florida
  - Research Site, Doral, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Homestead, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Albany, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Gurnee, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Quincy, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Northfield, New Jersey
  - Research Site, Union, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Hodges, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Arlington, Texas
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Splendora, Texas
  - Research Site, Provo, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Abingdon, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Greenfield, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (15):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Concepción del Uruguay
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, Godoy Cruz
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Nueve de Julio
  - Research Site, Ranelagh
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Australia (11):
  - Research Site, Bedford Park
  - Research Site, Box Hill
  - Research Site, Clayton
  - Research Site, Concord
  - Research Site, Frankston
  - Research Site, Nedlands
  - Research Site, New Lambton Heights
  - Research Site, Parkville
  - Research Site, Prahran
  - Research Site, Randwick
  - Research Site, Woolloongabba
- Brazil (4):
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Bulgaria (14):
  - Research Site, Dupnitsa
  - Research Site, Pazardzhik
  - Research Site, Pernik
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Samokov
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Velingrad
  - Research Site, Vratsa
  - Research Site, Yambol
- Canada (9):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
- Chile (5):
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Valparaíso
  - Research Site, Viña del Mar
- Czechia (8):
  - Research Site, Jindřichův Hradec
  - Research Site, Karlovy Vary
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Strakonice
  - Research Site, Teplice
- France (13):
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Mans
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pringy
  - Research Site, Saint-Pierre
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (18):
  - Research Site, Aschaffenburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Geesthacht
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Herford
  - Research Site, Leipzig
  - Research Site, Mainz Am Rhein
  - Research Site, München
  - Research Site, Neu-Isenburg
  - Research Site, Rostock
  - Research Site, Rüdersdorf
  - Research Site, Witten
- Japan (30):
  - Research Site, Asahi-shi
  - Research Site, Chiyoda-ku
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Itabashi-ku
  - Research Site, Kagoshima
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Kokubunji-shi
  - Research Site, Matsue
  - Research Site, Minatoku
  - Research Site, Mizunami-shi
  - Research Site, Niigata
  - Research Site, Obihiro-shi
  - Research Site, Ota-shi
  - Research Site, Ōita
  - Research Site, Sagamihara-shi
  - Research Site, Sakaide-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Setagaya-ku
  - Research Site, Shibuya-ku
  - Research Site, Shinagawa-ku
  - Research Site, Sumida-ku
  - Research Site, Takamatsu
  - Research Site, Toshima-ku
  - Research Site, Tsukubo-gun
  - Research Site, Yokohama
- Peru (2):
  - Research Site, Cusco
  - Research Site, Lima
- Philippines (3):
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Quezon City
- Poland (33):
  - Research Site, Aleksandrów Łódzki
  - Research Site, Bialystok
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Bystra
  - Research Site, Dobre Miasto
  - Research Site, Gdansk
  - Research Site, Giżycko
  - Research Site, Gorzów Wlkp
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Karczew
  - Research Site, Katowice
  - Research Site, Koszalin
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Lublin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Poznan
  - Research Site, Proszowice
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Skierniewice
  - Research Site, Sosnowiec
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Trzebnica
  - Research Site, Warsaw
  - Research Site, Wieluń
  - Research Site, Wołomin
  - Research Site, Wroclaw
  - Research Site, Żnin
- Romania (5):
  - Research Site, Bragadiru
  - Research Site, Bucharest
  - Research Site, Constanța
  - Research Site, Deva
  - Research Site, Iași
- Russia (18):
  - Research Site, Chelyabinsk
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, StPetersburg
  - Research Site, Tomsk
  - Research Site, Vladikavkaz
  - Research Site, Vladimir
  - Research Site, Volgograd
  - Research Site, Yekaterinburg
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, KwaDukuza
  - Research Site, Mowbray
- South Korea (9):
  - Research Site, Anyang-si
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Jeju City
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Sagunto(Valencia)
  - Research Site, Salamanca
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Lund
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Mersin
- Ukraine (8):
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (17):
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Cambridge
  - Research Site, Chertsey
  - Research Site, Chester
  - Research Site, Cottingham
  - Research Site, Darlington
  - Research Site, Glasgow
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Portsmouth
  - Research Site, Soham
  - Research Site, Somerset
  - Research Site, Stevenage
  - Research Site, Stockton
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Busse WW, Bleecker ER, FitzGerald JM, Ferguson GT, Barker P, Brooks L, Olsson RF, Martin UJ, Goldman M; BORA study investigators. Benralizumab for adolescent patients with severe, eosinophilic asthma: Safety and efficacy after 3 years of treatment. J Allergy Clin Immunol. 2021 Jul;148(1):266-271.e2. doi: 10.1016/j.jaci.2021.02.009. Epub 2021 Feb 17. PMID 33609624
- [Derived] Busse WW, Bleecker ER, FitzGerald JM, Ferguson GT, Barker P, Sproule S, Olsson RF, Martin UJ, Goldman M; BORA study investigators. Long-term safety and efficacy of benralizumab in patients with severe, uncontrolled asthma: 1-year results from the BORA phase 3 extension trial. Lancet Respir Med. 2019 Jan;7(1):46-59. doi: 10.1016/S2213-2600(18)30406-5. Epub 2018 Nov 8. PMID 30416083
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2560&filename=D3250C00021_Revised_CSP_3_16Dec2016_Redacted.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2560&filename=D3250C00021_SAP_Edition_3_11_Dec2017_Redacted.pdf
- See also: BORA clinical study protocol-redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2560&filename=BORA_clinical_study_protocol-redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2133 patients entered BORA. 10 were excluded due to a GCP breach. Of remaining 2123 patients, 1926 entered from SIROCCO/CALIMA and 197 from ZONDA. 2 patients were not treated, and a total of 447 patients (348 SIROCCO/CALIMA and 99 ZONDA) were later enrolled into MELTEMI without completing the follow-up in BORA, so not in the main analyses.
Pre-assignment Details: 953 participants from SIROCCO/CALIMA receive benralizumab 30 mg at every 4 weeks during BORA. 971 participants from SIROCCO/CALIMA receive treatment at every 8 weeks during BORA. 100 participants from ZONDA receive treatment at every 4 weeks during BORA. 97 participants from study ZONDA receive treatment at every 8 weeks during BORA.
Groups:
- SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks; ZONDA - Benralizumab 30 mg q.4 Weeks: Benralizumab administered subcutaneously every 4 weeks
- SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks; ZONDA - Benralizumab 30 mg q.8 Weeks: Benralizumab administered subcutaneously every 8 weeks
Period: Overall Study
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Started | 953 | 973 | 100 | 97
Treated | 953 | 971 | 100 | 97
Adolescents Only | 25 | 61 | 0 | 0
Completed (Include patients enrolled into study MELTEMI (study 37)) | 911 (170 enrolled into study MELTEMI) | 924 (178 enrolled into study MELTEMI) | 92 (51 enrolled into study MELTEMI) | 92 (48 enrolled into study MELTEMI)
Not Completed | 42 | 49 | 8 | 5
Not completed — eg. not made to the visit | 7 | 4 | 0 | 1
Not completed — study specific discount. criteria | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 20 | 20 | 7 | 1
Not completed — Lost to Follow-up | 5 | 12 | 1 | 2
Not completed — Death | 5 | 4 | 0 | 1
Not completed — Adverse Event | 3 | 4 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0
Not completed — Eligibility criteria not fulfilled | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis population defined as treated for at least 1 treatment, excluding patients enrolled in MELTEMI.
Groups:
- Total: Total of all reporting groups
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 783 | 793 | 49 | 49 | 1674
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Full analysis set, excluding MELTEMI patients
  Years | 51.1 (13.79) | 48.9 (15.53) | 49.7 (10.35) | 52.7 (8.90) | 50.1 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set, exclude MELTEMI patients
  Participants
    Female | 503 | 470 | 27 | 29 | 1029
    Male | 280 | 323 | 22 | 20 | 645
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full analysis set
  Participants
    White | 599 | 612 | 45 | 42 | 1298
    Black and African American | 16 | 19 | 0 | 1 | 36
    Asian | 138 | 136 | 4 | 6 | 284
    Other | 30 | 26 | 0 | 0 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Basophils, Full Analysis Set, Excluding MELTEMI Patients
Description: Change from baseline in hematologic lab parameter of Basophils.
Time Frame: Week 56
Population: Full analysis set, excluding MELTEMI patients. For each lab tests, number of patients is the number of patients with available change from baseline value.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 691 | 703 | 39 | 42
10^9 cells/L | -0.005 (0.0223) | -0.005 (0.0239) | -0.007 (0.0283) | -0.005 (0.0244)

2. Primary Outcome: Change From Baseline in Basophils, Full Analysis Set, Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline in hematologic lab parameter of Basophils.
Time Frame: Week 108
Population: Full analysis set, adolescents only (studies SIROCCO/CALIMA only, study ZONDA does not enroll adolescents). For each lab tests, number of patients is the number of patients with available change from baseline value.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 16 | 45
10^9 cells/L | -0.006 (0.0145) | 0.001 (0.0208)

3. Primary Outcome: Change From Baseline in Leukocytes, Full Analysis Set, Excluding MELTEMI Patients
Description: Change from baseline in hematologic lab parameter of Leukocytes.
Time Frame: Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 695 | 710 | 39 | 42
10^9 cells/L | -0.344 (2.0412) | -0.128 (1.8614) | -0.808 (1.8177) | -0.507 (3.3612)

4. Primary Outcome: Change From Baseline in Leukocytes, Full Analysis Set, Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline in hematologic lab parameter of Leukocytes.
Time Frame: Week 108
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 16 | 47
10^9 cells/L | -0.487 (1.7289) | -0.079 (1.8432)

5. Primary Outcome: Change From Baseline in Lymphocytes, Full Analysis Set, Excluding MELTEMI Patients
Description: Change from baseline in hematologic lab parameter of Lymphocytes.
Time Frame: Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 691 | 703 | 39 | 42
10^9 cells/L | -0.032 (0.6242) | 0.003 (0.5402) | -0.093 (0.6403) | 0.007 (0.6864)

6. Primary Outcome: Change From Baseline in Lymphocytes, Full Analysis Set, Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline in hematologic lab parameter of Lymphocytes.
Time Frame: Week 108
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 16 | 45
10^9 cells/L | -0.180 (0.6946) | -0.070 (0.6671)

7. Primary Outcome: Change From Baseline in Neutrophils, Full Analysis Set, Excluding MELTEMI Patients
Description: Change from baseline in hematologic lab parameter of Neutrophils.
Time Frame: Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 691 | 703 | 39 | 42
10^9 cells/L | -0.171 (1.8746) | 0.013 (1.7024) | -0.501 (1.7096) | -0.368 (3.2057)

8. Primary Outcome: Change From Baseline in Neutrophils, Full Analysis Set, Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline in hematologic lab parameter of Neutrophils.
Time Frame: Week 108
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 16 | 45
10^9 cells/L | -0.451 (1.7645) | 0.242 (1.8469)

9. Primary Outcome: Change From Baseline in Eosinophils, Full Analysis Set, Excluding MELTEMI Patients
Description: Change from baseline in hematologic lab parameter of Eosinophils.
Time Frame: Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 691 | 703 | 39 | 42
10^9 cells/L | -0.1220 (0.30599) | -0.1271 (0.26161) | -0.1451 (0.30766) | -0.1664 (0.35139)

10. Primary Outcome: Change From Baseline in Eosinophils, Full Analysis Set, Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline in hematologic lab parameter of Eosinophils.
Time Frame: Week 108
Population: Full analysis set, adolescents only(studies SIROCCO/CALIMA only, study ZONDA does not enroll adolescents). For each lab tests, number of patients is the number of patients with available change from baseline value.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 16 | 45
10^9 cells/L | -0.1294 (0.27973) | -0.1838 (0.3381)

11. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Full Analysis Set, Excluding MELTEMI Patients
Description: Change from baseline in chemistry tests ALT.
Time Frame: Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 684 | 712 | 37 | 43
ukat/L | -0.007 (0.2102) | 0.017 (0.4651) | -0.064 (0.3547) | -0.023 (0.1940)

12. Primary Outcome: Change From Baseline in ALT, Full Analysis Set, Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline in hematologic lab parameter of ALT.
Time Frame: Week 108
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 17 | 51
ukat/L | 0.048 (0.2195) | 0.034 (0.2312)

13. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Full Analysis Set, Excluding MELTEMI Patients
Description: Change from baseline in chemistry tests AST.
Time Frame: Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 684 | 712 | 37 | 43
ukat/L | -0.005 (0.1431) | 0.004 (0.3303) | -0.027 (0.2291) | -0.026 (0.1178)

14. Primary Outcome: Change From Baseline in AST, Full Analysis Set, Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline in hematologic lab parameter of AST.
Time Frame: Week 108
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 17 | 50
ukat/L | -0.006 (0.1196) | -0.013 (0.1297)

15. Primary Outcome: Change From Baseline in Bilirubin, Full Analysis Set, Excluding MELTEMI Patients
Description: Change from baseline in chemistry test Bilirubin.
Time Frame: Week 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 685 | 712 | 37 | 43
umol/L | 0.187 (3.6261) | 0.391 (3.9945) | 0.146 (2.8094) | 0.279 (3.8765)

16. Primary Outcome: Change From Baseline in Bilirubin, Full Analysis Set, Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline in hematologic lab parameter of Bilirubin.
Time Frame: Week 108
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 17 | 51
umol/L | 2.221 (8.3453) | 0.202 (3.6575)

17. Secondary Outcome: Number of Overall Patients With Asthma Exacerbations During Study Period
Description: Annual asthma exacerbation rate, where an asthma exacerbation is defined by a worsening of asthma requiring the use of systemic corticosteroids for at least 3 days, and/or an in patient hospitalization, and/or an emergency department or urgent care visit
Time Frame: From week 0 to week 56 in study treatment period and through the follow up period (16 weeks from day of last dose)
Population: Full analysis set, excluding MELTEMI patients. Summarized by subsets of patients enrolled from SIROCCO/CALIMA with baseline eosinophils count >=300/uL or <300/uL; all patients enrolled from ZONDA; separated by predecessor treatment groups.
Measure: Count of Participants; unit: Participants
Groups:
- SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4; ZONDA - Benralizumab 30 mg q.4 - Pre Benra q.4: Benralizumab administered subcutaneously every 4 weeks, predecessor study with benralizumab treatment
- SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo; ZONDA - Benralizumab 30 mg q.4 - Predecessor Placebo: Benralizumab administered subcutaneously every 4 weeks, predecessor study with placebo treatment
- SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8; ZONDA - Benralizumab 30 mg q.8 - Pre Benra q.8: Benralizumab administered subcutaneously every 8 weeks, predecessor study with benralizumab treatment
- SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo; ZONDA - Benralizumab 30 mg q.8 - Predecessor Placebo: Benralizumab administered subcutaneously every 8 weeks, predecessor study with placebo treatment
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 - Pre Benra q.4 | ZONDA - Benralizumab 30 mg q.4 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 - Pre Benra q.8 | ZONDA - Benralizumab 30 mg q.8 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 518 | 265 | 783 | 512 | 281 | 793 | 31 | 18 | 49 | 31 | 18 | 49
Participants
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 347 | 172 | 519 | 339 | 188 | 527 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL: Number of exacerbation | 99 | 60 | 159 | 104 | 66 | 170 |  |  |  |  |  |
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 171 | 93 | 264 | 173 | 93 | 266 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos<300/μL: Number of exacerbation | 69 | 44 | 113 | 65 | 32 | 97 |  |  |  |  |  |
  Zonda Patients with asthma exacerbations: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 18 | 49 | 31 | 18 | 49
  Zonda Patients with asthma exacerbations: Number of exacerbation |  |  |  |  |  |  | 12 | 5 | 17 | 13 | 11 | 24

18. Secondary Outcome: Number of Overall Patients With Asthma Exacerbations During Study Period, Adolescents Only (SIROCCO/CALIMA)
Description: as for outcome 17
Time Frame: From week 0 to week 108 in study treatment period and through the follow up period (16 weeks from day of last dose)
Population: Full analysis set, adolescents only (studies SIROCCO/CALIMA only, study ZONDA does not enroll adolescents). Summarized by subsets of patients enrolled from SIROCCO/CALIMA with baseline eosinophils count >=300/uL or <300/uL; separated by predecessor treatment groups.
Measure: Count of Participants; unit: Participants
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 14 | 11 | 25 | 32 | 29 | 61
Participants
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 11 | 9 | 20 | 17 | 14 | 31
  Sirocco/Calima patients with eos>=300/μL: Number of exacerbation | 2 | 6 | 8 | 3 | 5 | 8
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 3 | 2 | 5 | 15 | 15 | 30
  Sirocco/Calima patients with eos<300/μL: Number of exacerbation | 0 | 0 | 0 | 5 | 6 | 11

19. Secondary Outcome: Change From Baseline in Pre-bronchodilator FEV1 (L)
Description: Change from baseline to Week 56 in Pre-bronchodilator Forced expiratory volume in 1 second (FEV1).
Time Frame: Week 56
Population: Full analysis set, excluding MELTEMI patients. For patients enrolled from SIROCCO/CALIMA, summarized by baseline eosinophils count>=300/uL, and <300/uL; all patients enrolled from ZONDA; separated by predecessor treatment groups.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 - Pre Benra q.4 | ZONDA - Benralizumab 30 mg q.4 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 - Pre Benra q.8 | ZONDA - Benralizumab 30 mg q.8 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 444 | 221 | 665 | 440 | 220 | 660 | 31 | 18 | 38 | 28 | 15 | 43
L
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 297 | 142 | 439 | 291 | 151 | 442 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL | -0.006 (0.295) | 0.131 (0.422) | 0.038 (0.346) | 0.019 (0.317) | 0.081 (0.419) | 0.040 (0.356) |  |  |  |  |  |
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 147 | 79 | 226 | 149 | 69 | 218 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos<300/μL | -0.021 (0.376) | -0.011 (0.280) | -0.017 (0.345) | -0.015 (0.293) | 0.030 (0.350) | -0.001 (0.312) |  |  |  |  |  |
  Number of Zonda Patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 18 | 38 | 28 | 15 | 43
  Number of Zonda Patients |  |  |  |  |  |  | 0.013 (0.354) | 0.167 (0.533) | 0.057 (0.412) | -0.093 (0.280) | 0.138 (0.329) | -0.012 (0.314)

20. Secondary Outcome: Change From Baseline in Pre-bronchodilator FEV1 (L), Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline to Week 108 in Pre-bronchodilator Forced expiratory volume in 1 second (FEV1).
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 8 | 9 | 17 | 25 | 26 | 51
L
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 6 | 8 | 14 | 13 | 13 | 26
  Sirocco/Calima patients with eos>=300/μL | 0.205 (0.289) | -0.189 (0.354) | -0.020 (0.375) | 0.578 (0.608) | 0.413 (0.375) | 0.496 (0.502)
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 2 | 1 | 3 | 12 | 13 | 25
  Sirocco/Calima patients with eos<300/μL | 0.325 (0.431) | 1.140 (NA) — Only 1 participants, not able to calculate Standard deviation. | 0.597 (0.561) | 0.047 (0.340) | 0.240 (0.519) | 0.147 (0.444)

21. Secondary Outcome: Change From Baseline in Post-bronchodilator FEV1 (L)
Description: Change from baseline to Week 56 in Post-bronchodilator Forced expiratory volume in 1 second (FEV1).
Time Frame: Week 56
Population: Full analysis set, excluding MELTEMI patients. Only summarize for patients enrolled from SIROCCO/CALIMA, summarized by baseline eosinophils count>=300/uL, and <300/uL; separated by predecessor treatment groups. Patients from Study ZONDA are not summarized.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 439 | 220 | 659 | 438 | 214 | 652
L
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 296 | 144 | 440 | 292 | 151 | 443
  Sirocco/Calima patients with eos>=300/μL | -0.066 (0.280) | 0.089 (0.455) | -0.015 (0.354) | -0.029 (0.281) | 0.045 (0.401) | -0.004 (0.329)
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 143 | 76 | 219 | 146 | 63 | 209
  Sirocco/Calima patients with eos<300/μL | -0.058 (0.379) | -0.024 (0.289) | -0.046 (0.350) | -0.043 (0.273) | 0.049 (0.394) | -0.015 (0.316)

22. Secondary Outcome: Change From Baseline in Post-bronchodilator FEV1 (L), Adolescents Only (SIROCCO/CALIMA)
Description: Change from baseline to Week 108 in Post-bronchodilator Forced expiratory volume in 1 second (FEV1).
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 8 | 9 | 17 | 25 | 26 | 51
L
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 6 | 8 | 14 | 13 | 13 | 26
  Sirocco/Calima patients with eos>=300/μL | -0.062 (0.537) | -0.305 (0.394) | -0.201 (0.458) | 0.603 (0.749) | 0.279 (0.659) | 0.448 (0.712)
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 2 | 1 | 3 | 12 | 13 | 25
  Sirocco/Calima patients with eos<300/μL | 0.375 (0.474) | 0.880 (NA) — Only 1 participants, not able to calculate SD | 0.543 (0.444) | -0.006 (0.327) | 0.218 (0.536) | 0.111 (0.454)

23. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) as a Measure of Asthma Control in Overall Patients
Description: Asthma Control Questionnaire 6 (ACQ-6) contains 1 bronchodilator use question and 5 symptom questions. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-6 score was the mean of the responses.
Time Frame: Week 56
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 - Pre Benra q.4 | ZONDA - Benralizumab 30 mg q.4 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 - Pre Benra q.8 | ZONDA - Benralizumab 30 mg q.8 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 447 | 224 | 671 | 444 | 220 | 664 | 28 | 11 | 39 | 28 | 15 | 43
Score on a scale
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 298 | 146 | 444 | 294 | 153 | 447 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL | -0.04 (0.83) | -0.20 (1.04) | -0.09 (0.91) | -0.06 (0.82) | -0.25 (1.06) | -0.12 (0.91) |  |  |  |  |  |
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 149 | 78 | 227 | 150 | 67 | 217 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos<300/μL | -0.16 (0.90) | -0.12 (0.80) | -0.15 (0.86) | -0.10 (0.83) | -0.09 (1.06) | -0.10 (0.90) |  |  |  |  |  |
  Number of Zonda Patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 11 | 39 | 28 | 15 | 43
  Number of Zonda Patients |  |  |  |  |  |  | -0.05 (0.89) | -0.61 (0.74) | -0.21 (0.87) | 0.15 (1.02) | -0.43 (1.00) | -0.05 (1.04)

24. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) as a Measure of Asthma Control in Overall Patients, Adolescents Only (SIROCCO/CALIMA)
Description: as for outcome 23
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 9 | 9 | 18 | 25 | 26 | 51
Score on a scale
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 7 | 8 | 15 | 13 | 13 | 26
  Sirocco/Calima patients with eos>=300/μL | 0.26 (0.53) | 0.06 (0.49) | 0.16 (0.50) | -0.14 (0.51) | -0.10 (1.38) | -0.12 (1.02)
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 2 | 1 | 3 | 12 | 13 | 25
  Sirocco/Calima patients with eos<300/μL | -0.50 (0.24) | -1.83 (NA) — Only one participant, not able to calculate SD. | 0.94 (0.79) | -0.21 (0.78) | -0.21 (0.77) | -0.21 (0.76)

25. Secondary Outcome: Change From Baseline in Total Score of Asthma Related and General Health-related Quality of Life Questionnaire (AQLQ(S)+12)
Description: Standardised Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(S)+12) comprises 4 separate domains (symptoms, activity limitations, emotional function, and environmental stimuli). It contains 32 questions on a 7 point scale ranging from 7 (no impairment) to 1 (severe impairment); total score is an average of all questions. An increase in score indicates improvement.
Time Frame: Week 56
Population: Full analysis set, excluding MELTEMI patients. For patients enrolled from SIROCCO/CALIMA, summarized by baseline eosinophils count>=300/uL, and <300/uL; all patients enrolled from ZONDA.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 - Pre Benra q.4 | ZONDA - Benralizumab 30 mg q.4 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 - Pre Benra q.8 | ZONDA - Benralizumab 30 mg q.8 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 444 | 224 | 668 | 442 | 220 | 662 | 26 | 11 | 37 | 28 | 15 | 43
Score on a scale
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 296 | 146 | 442 | 293 | 153 | 446 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL | 0.02 (0.80) | 0.21 (0.98) | 0.08 (0.87) | 0.08 (0.91) | 0.26 (1.00) | 0.15 (0.94) |  |  |  |  |  |
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 148 | 78 | 226 | 149 | 67 | 216 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos<300/μL | 0.11 (0.84) | 0.03 (0.89) | 0.09 (0.85) | 0.15 (0.90) | 0.02 (1.06) | 0.11 (0.95) |  |  |  |  |  |
  Number of Zonda Patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 11 | 37 | 28 | 15 | 43
  Number of Zonda Patients |  |  |  |  |  |  | 0.13 (0.93) | 0.43 (0.91) | 0.22 (0.92) | -0.04 (0.94) | 0.40 (1.03) | 0.11 (0.98)

26. Secondary Outcome: Change From Baseline in Total Score of Asthma Related and General Health-related Quality of Life Questionnaire (AQLQ(S)+12), Adolescents Only (SIROCCO/CALIMA)
Description: as for outcome 25
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 9 | 8 | 17 | 25 | 26 | 51
Score on a scale
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 7 | 7 | 14 | 13 | 13 | 26
  Sirocco/Calima patients with eos>=300/μL | 0.60 (1.22) | -0.11 (0.21) | 0.25 (0.92) | 0.52 (0.37) | 0.06 (0.59) | 0.29 (0.54)
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 2 | 1 | 3 | 12 | 13 | 25
  Sirocco/Calima patients with eos<300/μL | 0.64 (0.55) | 1.53 (NA) — Only one participants, not able to calculate SD. | 0.94 (0.65) | 0.58 (1.01) | 0.27 (0.77) | 0.42 (0.89)

27. Secondary Outcome: Change of Blood Eosinophil Levels' Measurement in Overall Patients
Description: Change from baseline to Week 56 in Blood eosinophils
Time Frame: Week 56
Population: Full analysis set, excluding MELTEMI patients. For patients enrolled from SIROCCO/CALIMA, summarized by baseline eosinophils count>=300/uL, and <300/uL; all patients enrolled from ZONDA; separate by predecessor treatment groups.
Measure: Mean (Standard Deviation); unit: cell/uL
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 - Pre Benra q.4 | ZONDA - Benralizumab 30 mg q.4 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 - Pre Benra q.8 | ZONDA - Benralizumab 30 mg q.8 - Predecessor Placebo | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 454 | 237 | 691 | 461 | 242 | 703 | 28 | 11 | 39 | 27 | 15 | 42
cell/uL
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 306 | 156 | 462 | 302 | 162 | 464 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL | 4.9 (177.42) | -449.6 (360.6) | -148.6 (332.91) | -10.1 (134.7) | -422.5 (330.01) | -154.1 (297.34) |  |  |  |  |  |
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 148 | 81 | 229 | 159 | 80 | 239 | 0 | 0 | 0 | 0 | 0 | 0
  Sirocco/Calima patients with eos<300/μL | 15.7 (87.04) | -222.1 (325.03) | -68.4 (234.40) | -2.9 (59.11) | -217.4 (198.56) | -74.7 (160.29) |  |  |  |  |  |
  Number of Zonda Patients: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 11 | 39 | 27 | 15 | 42
  Number of Zonda Patients |  |  |  |  |  |  | 2.5 (69.85) | -520.9 (360.79) | -145.1 (307.66) | -17.0 (107.48) | -435.3 (468.64) | -166.4 (351.39)

28. Secondary Outcome: Change of Blood Eosinophil Levels' Measurement in Adolescents Patients (SIROCCO/CALIMA).
Description: Change from baseline to Week 108 in Blood eosinophils.
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: cell/uL
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 7 | 7 | 14 | 21 | 16 | 37
cell/uL
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 6 | 6 | 12 | 11 | 7 | 18
  Sirocco/Calima patients with eos>=300/μL | 78.3 (192.19) | -356.7 (215.47) | -139.2 (299.16) | -163.6 (502.76) | -332.9 (349.89) | -229.4 (446.21)
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 1 | 1 | 2 | 10 | 9 | 19
  Sirocco/Calima patients with eos<300/μL | 160.0 (NA) — Only one participants, not able to calculate SD. | -150.0 (NA) — Only one participants, not able to calculate SD. | 5.0 (219.20) | -2.0 (9.19) | -204.4 (152.32) | -97.9 (145.40)

29. Secondary Outcome: Change From Baseline in EQ-5D-5L Visual Analog Scale
Description: The questionnaire included a visual analog scale (VAS) score, where the patient was asked to rate current health status on a scale of 0 to 100, with 0 being the worst imaginable health state; thus, an increase in VAS score indicated improvement.
Time Frame: Week 56
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 682 | 709 | 21 | 28
Score on a scale
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 454 | 468 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL | 6.08 (15.68) | 6.02 (17.68) |  |
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 228 | 241 | 0 | 0
  Sirocco/Calima patients with eos<300/μL | 4.38 (14.99) | 6.69 (15.96) |  |
  Number of Zonda Patients: number analyzed (Participants) | 0 | 0 | 21 | 28
  Number of Zonda Patients |  |  | 5.00 (10.35) | 1.36 (13.58)

30. Secondary Outcome: Change From Baseline in EQ-5D-5L Visual Analog Scale, Adolescents Only (SIROCCO/CALIMA)
Description: The questionnaire included a VAS, where the patient was asked to rate current health status on a scale of 0 to 100, with 0 being the worst imaginable health state; thus, an increase in VAS score indicated improvement.
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 9 | 9 | 18 | 24 | 24 | 48
Score on a scale
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 7 | 8 | 15 | 13 | 12 | 25
  Sirocco/Calima patients with eos>=300/μL | 5.43 (9.73) | 6.63 (15.53) | 6.07 (12.71) | 11.54 (26.95) | 9.83 (13.87) | 10.72 (21.26)
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 2 | 1 | 3 | 11 | 12 | 23
  Sirocco/Calima patients with eos<300/μL | 22.00 (12.73) | -4.00 (NA) — Only one participants, not able to calculate SD. | 13.33 (17.50) | 10.18 (32.69) | 5.08 (10.45) | 7.52 (23.39)

31. Secondary Outcome: Work Productivity Loss in Adults, Using Work Productivity and Activity Impairment Questionnaire (WPAI)
Description: The WPAI+CIQ is a 10-item questionnaire that assesses productivity and activity impairment over the previous week. The questionnaire includes hours missed from work/school due to asthma, degree health affected productivity while at work/school, as well as the degree to which health affected regular activities other than work or school. The questionnaire related to the previous 7 days. Work productivity loss is calculated with sum of hours missed at work due to health problem and hours that affected due to health problem at work, divided by sum of hours missed due to health problem and hours actually worked, presented by percentage.
Time Frame: Week 68
Population: Full analysis set, adults, excluding MELTEMI patients. Summarized by subsets of patients enrolled from SIROCCO/CALIMA with baseline eosinophils count >=300/uL or <300/uL; all patients enrolled from ZONDA.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 349 | 313 | 19 | 20
percentage
  Sirocco/Calima patients with eos>=300/μL-wk 68: number analyzed (Participants) | 236 | 217 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL-wk 68 | 23.3 (26.18) | 21.0 (25.54) |  |
  Sirocco/Calima patients with eos<300/μL-wk 68: number analyzed (Participants) | 113 | 96 | 0 | 0
  Sirocco/Calima patients with eos<300/μL-wk 68 | 32.7 (27.55) | 25.8 (24.05) |  |
  Zonda Patients-wk 68: number analyzed (Participants) | 0 | 0 | 19 | 20
  Zonda Patients-wk 68 |  |  | 18.9 (24.94) | 21.0 (27.13)

32. Secondary Outcome: Work Productivity Loss in Adults, Using Work Productivity and Activity Impairment Questionnaire (WPAI), Adolescents Only (SIROCCO/CALIMA)
Description: as for outcome 31
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 2 | 1 | 3 | 3 | 4 | 7
Percentage
  Sirocco/Calima patients with eos>=300/μL-wk 108: number analyzed (Participants) | 2 | 1 | 3 | 1 | 1 | 2
  Sirocco/Calima patients with eos>=300/μL-wk 108 | 0.0 (0.00) | 10.0 (NA) — Only one participant, not able to calculate SD. | 3 (3.3) | 20.0 (NA) — Only one participant, not able to calculate SD. | 10.0 (NA) — Only one participant, not able to calculate SD. | 15.0 (7.07)
  Sirocco/Calima patients with eos<300/μL-wk-108: number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 5
  Sirocco/Calima patients with eos<300/μL-wk-108 |  |  |  | 0.0 (0.00) | 13.3 (5.77) | 8.0 (8.37)

33. Secondary Outcome: Classroom Productivity Loss Using Classroom Impairment Questionnaire (CIQ)
Description: The WPAI (+CIQ) is a 10-item questionnaire that assesses productivity and activity impairment over the previous week. The questionnaire includes hours missed from work/school due to asthma, degree health affected productivity while at work/school, as well as the degree to which health affected regular activities other than work or school. The questionnaire related to the previous 7 days. Classroom productivity loss is calculated with sum of hours missed for classes due to health problem and hours that affected due to health problem in classes, divided by sum of hours missed due to health problem and hours actually attended classes, presented by percentage.
Time Frame: Week 56
Population: Full analysis set, adolescents, excluding MELTEMI patients. For patients enrolled from SIROCCO/CALIMA, summarized by baseline eosinophils count>=300/uL, and <300/uL; all patients enrolled from ZONDA.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 10 | 48 | 0 | 0
Percentage
  Sirocco/Calima patients with eos>=300/μL-wk 56: number analyzed (Participants) | 8 | 24 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL-wk 56 | 3.8 (7.44) | 15.2 (20.69) |  |
  Sirocco/Calima patients with eos<300/μL-wk 56: number analyzed (Participants) | 2 | 24 | 0 | 0
  Sirocco/Calima patients with eos<300/μL-wk 56 | 5.0 (7.07) | 17.1 (20.06) |  |
  Zonda patients-wk 56: number analyzed (Participants) | 0 | 0 | 0 | 0

34. Secondary Outcome: Classroom Productivity Loss Using Classroom Impairment Questionnaire (CIQ), Adolescents Only (SIROCCO/CALIMA)
Description: as for outcome 33
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 7 | 4 | 11 | 19 | 21 | 40
Percentage
  Sirocco/Calima patients with eos>=300/μL-wk 108: number analyzed (Participants) | 5 | 4 | 9 | 10 | 11 | 21
  Sirocco/Calima patients with eos>=300/μL-wk 108 | 4.9 (6.82) | 15.2 (17.55) | 9.5 (12.98) | 5.4 (8.32) | 18.6 (27.94) | 12.3 (21.62)
  Sirocco/Calima patients with eos<300/μL-wk-108: number analyzed (Participants) | 2 | 0 | 2 | 9 | 10 | 19
  Sirocco/Calima patients with eos<300/μL-wk-108 | 21.5 (30.41) |  | 21.5 (30.41) | 12.5 (18.10) | 10.6 (11.68) | 11.5 (14.66)

35. Secondary Outcome: Activity Impairment (%), Using Work Productivity and Activity Impairment Questionnaire (WPAI)
Description: The WPAI+CIQ is a 10-item questionnaire that assesses productivity and activity impairment over the previous week. The questionnaire includes hours missed from work/school due to asthma, degree health affected productivity while at work/school, as well as the degree to which health affected regular activities other than work or school. The questionnaire related to the previous 7 days. The WPAI+CIQ outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Week 68
Population: Full analysis set, excluding MELTEMI patients. Summarized by subsets of patients enrolled from SIROCCO/CALIMA with baseline eosinophils count >=300/uL or <300/uL; all patients enrolled from ZONDA.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 697 | 674 | 38 | 41
percentage
  Sirocco/Calima patients with eos>=300/μL-wk 68: number analyzed (Participants) | 458 | 454 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL-wk 68 | 26.6 (26.14) | 24.4 (25.26) |  |
  Sirocco/Calima patients with eos<300/μL-wk 68: number analyzed (Participants) | 239 | 220 | 0 | 0
  Sirocco/Calima patients with eos<300/μL-wk 68 | 33.6 (26.55) | 32.7 (26.58) |  |
  Zonda Patients-wk 68: number analyzed (Participants) | 0 | 0 | 38 | 41
  Zonda Patients-wk 68 |  |  | 28.4 (27.85) | 39.0 (34.36)

36. Secondary Outcome: Activity Impairment (%), Using Work Productivity and Activity Impairment Questionnaire (WPAI), Adolescents Only (SIROCCO/CALIMA)
Description: as for outcome 35
Time Frame: Week 108
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 9 | 9 | 18 | 25 | 26 | 50
Percentage
  Sirocco/Calima patients with eos>=300/μL-wk 108: number analyzed (Participants) | 7 | 8 | 15 | 13 | 13 | 26
  Sirocco/Calima patients with eos>=300/μL-wk 108 | 7.1 (11.13) | 5.0 (9.26) | 6.0 (9.86) | 5.4 (8.77) | 19.2 (24.31) | 12.3 (19.25)
  Sirocco/Calima patients with eos<300/μL-wk-108: number analyzed (Participants) | 2 | 1 | 3 | 12 | 13 | 24
  Sirocco/Calima patients with eos<300/μL-wk-108 | 10.0 (14.14) | 20.0 (NA) — Only one participant, not able to calculate SD. | 13.3 (11.55) | 14.2 (18.81) | 11.5 (10.68) | 12.8 (14.87)

37. Secondary Outcome: Number of Patients Who Had Health Care Encounter (ie, Hospitalization, Emergency Department Visits, Urgent Care Visits, and All Other Outpatient Visits Due to Asthma) During Study Period
Description: Hospitalizations, Emergency department (ED) visits, urgent care visits and all other outpatient visits due to asthma
Time Frame: From week 0 to week 68 in study treatment period and through the follow up period (16 weeks from day of last dose)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 783 | 793 | 49 | 49
Participants
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 519 | 527 | 0 | 0
  Sirocco/Calima patients with eos>=300/μL | 193 | 198 |  |
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 264 | 266 | 0 | 0
  Sirocco/Calima patients with eos<300/μL | 118 | 102 |  |
  Number of Zonda Patients: number analyzed (Participants) | 0 | 0 | 49 | 49
  Number of Zonda Patients |  |  | 20 | 25

38. Secondary Outcome: Number of Patients Who Had Health Care Encounter (ie, Hospitalization, Emergency Department Visits, Urgent Care Visits, and All Other Outpatient Visits Due to Asthma) During Study Period, Adolescents Only (SIROCCO/CALIMA)
Description: Hospitalizations, ED visits, urgent care visits and all other outpatient visits due to asthma
Time Frame: Baseline and Week 108
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 14 | 11 | 25 | 32 | 29 | 61
Participants
  Sirocco/Calima patients with eos>=300/μL: number analyzed (Participants) | 11 | 9 | 20 | 17 | 14 | 31
  Sirocco/Calima patients with eos>=300/μL | 2 | 5 | 7 | 7 | 7 | 14
  Sirocco/Calima patients with eos<300/μL: number analyzed (Participants) | 3 | 2 | 5 | 15 | 15 | 30
  Sirocco/Calima patients with eos<300/μL | 0 | 1 | 1 | 7 | 5 | 12

39. Secondary Outcome: Pre-dose Benralizumab Concentration in Serum During the Treatment Phase of the Safety Study
Description: Endpoint: Pharmacokinetic (PK) parameters
Time Frame: Week 0 and Week 56
Population: All patients who received benralizumab, from whom PK blood samples were assumed not to be affected by factors such as protocol violations, and who had at least 1 quantifiable serum PK observation post the first dose were included in the PK analysis dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- ZONDA - Benra 30 mg q.4 Weeks - Pre Benra q.4: Benralizumab administered subcutaneously every 4 weeks, predecessor study with benralizumab treatment
- ZONDA - Benra 30 mg q.4 wk - Predecessor Placebo: Benralizumab administered subcutaneously every 4 weeks, predecessor study with placebo treatment
- ZONDA - Benra 30 mg q.8 Weeks - Pre Benra q.8: Benralizumab administered subcutaneously every 8 weeks, predecessor study with benralizumab treatment
- ZONDA - Benra 30 mg q.8 wk - Predecessor Placebo: Benralizumab administered subcutaneously every 8 weeks, predecessor study with placebo treatment
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo | ZONDA - Benra 30 mg q.4 Weeks - Pre Benra q.4 | ZONDA - Benra 30 mg q.4 wk - Predecessor Placebo | ZONDA - Benra 30 mg q.8 Weeks - Pre Benra q.8 | ZONDA - Benra 30 mg q.8 wk - Predecessor Placebo
Number analyzed (Participants) | 514 | 263 | 511 | 279 | 31 | 16 | 31 | 17
ng/mL
  Baseline: number analyzed (Participants) | 507 | 260 | 503 | 275 | 31 | 16 | 30 | 17
  Baseline | 714.25 [624.48 to 816.93] | NA [NA to NA] — Concentration <LLOQ (Lower Limit of Quantification) | 142.92 [124.08 to 164.63] | NA [NA to NA] — Concentration <LLOQ | 964.21 [589.87 to 1576.11] | NA [NA to NA] — Concentration <LLOQ | 692.91 [428.49 to 1120.50] | NA [NA to NA] — Concentration <LLOQ
  Week 56: number analyzed (Participants) | 442 | 225 | 440 | 215 | 27 | 10 | 27 | 15
  Week 56 | 930.04 [825.89 to 1047.33] | 865.93 [721.50 to 1039.27] | 173.95 [151.81 to 199.33] | 162.03 [132.31 to 195.43] | 823.62 [476.98 to 1422.17] | 1160.58 [833.77 to 1615.49] | 247.26 [165.87 to 368.57] | 139.35 [61.90 to 313.70]

40. Secondary Outcome: Pre-dose Benralizumab Concentration in Serum During the Treatment Phase of the Safety Study, Adolescents Only (SIROCCO/CALIMA)
Description: Endpoint: Pharmacokinetic (PK) parameters
Time Frame: Baseline and Week 108
Population: All adolescent patients (studies SIROCCO/CALIMA only, study ZONDA does not enroll adolescents)who received benralizumab, from whom PK blood samples were assumed not to be affected by factors such as protocol violations, and who had at least 1 quantifiable serum PK observation post the first dose were included in the PK analysis dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Pre Benra q.4 | SIROCCO/CALIMA - Benralizumab 30 mg q.4 - Predecessor Placebo | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Pre Benra q.8 | SIROCCO/CALIMA - Benralizumab 30 mg q.8 - Predecessor Placebo
Number analyzed (Participants) | 14 | 11 | 32 | 29
ng/mL
  Baseline: number analyzed (Participants) | 13 | 10 | 31 | 29
  Baseline | 725.55 [231.38 to 2275.13] | NA [NA to NA] — PK concentration <LLOQ (Lower limit of quantification) | 218.53 [126.53 to 377.42] | NA [NA to NA] — PK concentration <LLOQ
  Week 108: number analyzed (Participants) | 8 | 9 | 25 | 26
  Week 108 | 383.73 [30.90 to 4764.79] | 853.51 [260.26 to 2799.03] | 436.85 [185.36 to 1029.59] | 524.39 [287.72 to 955.74]

41. Secondary Outcome: Number of Patients With Anti-drug Antibodies (ADA) Responses During the Study
Description: Assessments for the presence of ADA and neutralizing antibody (nAb) throughout study
Time Frame: From week 0 to week 56 in study treatment period (adults) and plus 16 weeks the follow up period; From week 0 to week 108-week in study treatment period (adolescents) and plus 16 weeks the follow up period
Population: Full analysis set, excluding MELTEMI patients.
Measure: Number; unit: Participants
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 783 | 793 | 49 | 49
Participants
  Positive at any visit | 80 | 93 | 4 | 8
  Base- and Post-baseline Positive: number analyzed (Participants) | 774 | 789 | 47 | 48
  Base- and Post-baseline Positive | 23 | 41 | 2 | 4
  Newly Persistently Positive: number analyzed (Participants) | 774 | 789 | 47 | 48
  Newly Persistently Positive | 28 | 34 | 1 | 3
  Stable persistently positive: number analyzed (Participants) | 774 | 789 | 47 | 48
  Stable persistently positive | 21 | 29 | 2 | 2
  Newly treatment-induced positive: number analyzed (Participants) | 774 | 789 | 47 | 48
  Newly treatment-induced positive | 38 | 41 | 2 | 2
  ADA treatment boosted positive: number analyzed (Participants) | 774 | 789 | 47 | 48
  ADA treatment boosted positive | 6 | 6 | 0 | 1
  Decreased in titre: number analyzed (Participants) | 774 | 789 | 47 | 48
  Decreased in titre | 17 | 9 | 2 | 1
  Only post-baseline positive: number analyzed (Participants) | 774 | 789 | 47 | 48
  Only post-baseline positive | 48 | 48 | 2 | 1
  ADA incidence: number analyzed (Participants) | 774 | 789 | 47 | 48
  ADA incidence | 44 | 47 | 2 | 3
  Transiently Positive: number analyzed (Participants) | 774 | 789 | 47 | 48
  Transiently Positive | 22 | 26 | 1 | 3
  Only baseline positive: number analyzed (Participants) | 774 | 793 | 49 | 49
  Only baseline positive | 9 | 4 | 0 | 0
  nAb positive | 57 | 75 | 3 | 4

42. Secondary Outcome: Number of Patients With Anti-drug Antibodies (ADA) Responses During the Study, Adolescents Only (SIROCCO/CALIMA)
Description: Assessments for the presence of ADA and nAb throughout study
Time Frame: From week 0 to week 108 study treatment period (adults) and plus 16 weeks the follow up period; From week 0 to week 108-week in study treatment period (adolescents) and plus 16 weeks the follow up period
Population: Full analysis set, adolescents only (studies SIROCCO/CALIMA only, study ZONDA does not enroll adolescents).
Measure: Number; unit: Participants
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks
Number analyzed (Participants) | 25 | 61
Participants
  Positive at any visit | 1 | 5
  Base- and Post-baseline Positive | 0 | 3
  Newly Persistently Positive | 0 | 2
  Stable persistently positive | 0 | 3
  Newly treatment-induced positive | 1 | 1
  ADA treatment boosted positive | 0 | 2
  Decreased in titre | 0 | 2
  Only post-baseline positive | 1 | 2
  ADA incidence | 1 | 3
  Transiently Positive | 1 | 0
  Only baseline positive | 0 | 0
  nAb positive | 1 | 5

ADVERSE EVENTS:
Time Frame: Adults completed 56 weeks of treatment period and 12 weeks follow-up period; and adolescents completed 108 weeks of treatment period and 12 weeks follow-up period.
Arm/Group | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks | ZONDA - Benralizumab 30 mg q.4 Weeks | ZONDA - Benralizumab 30 mg q.8 Weeks
All-Cause Mortality (participants affected / at risk) | 5/783 | 4/793 | 0/49 | 1/49
Serious Adverse Events (participants affected / at risk) | 102/783 | 94/793 | 10/49 | 9/49
Other Adverse Events (participants affected / at risk) | 415/783 | 409/793 | 33/49 | 38/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks (N=783) | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks (N=793) | ZONDA - Benralizumab 30 mg q.4 Weeks (N=49) | ZONDA - Benralizumab 30 mg q.8 Weeks (N=49)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Solid pseudopapillary tumour of the pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocrine test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 36 (40) | 26 (31) | 3 (4) | 2 (2)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle lobe syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIROCCO/CALIMA - Benralizumab 30 mg q.4 Weeks (N=783) | SIROCCO/CALIMA - Benralizumab 30 mg q.8 Weeks (N=793) | ZONDA - Benralizumab 30 mg q.4 Weeks (N=49) | ZONDA - Benralizumab 30 mg q.8 Weeks (N=49)
Influenza like illness (General disorders) | 27 (41) | 30 (35) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 50 (66) | 51 (76) | 3 (7) | 10 (16)
Upper respiratory tract infection (Infections and infestations) | 61 (95) | 56 (82) | 0 (0) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (32) | 20 (20) | 5 (5) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 4 (5) | 8 (8) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 9 (9) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 6 (6) | 7 (8) | 2 (2) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11) | 5 (13) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 4 (6) | 0 (0) | 2 (3)
Oedema peripheral (General disorders) | 4 (4) | 6 (7) | 0 (0) | 4 (6)
Seasonal allergy (Immune system disorders) | 13 (15) | 8 (8) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 27 (46) | 44 (61) | 2 (5) | 2 (4)
Bronchitis bacterial (Infections and infestations) | 19 (24) | 16 (22) | 3 (3) | 2 (2)
Chronic sinusitis (Infections and infestations) | 12 (13) | 10 (17) | 1 (1) | 2 (7)
Herpes zoster (Infections and infestations) | 8 (8) | 2 (2) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 14 (20) | 13 (16) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 24 (28) | 26 (37) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 8 (8) | 12 (13) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 22 (25) | 18 (22) | 3 (3) | 4 (4)
Upper respiratory tract infection bacterial (Infections and infestations) | 15 (17) | 23 (28) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 14 (17) | 8 (8) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 124 (186) | 130 (196) | 14 (22) | 13 (19)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 4 (5) | 3 (3) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (25) | 21 (21) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 38 (54) | 40 (55) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 12 (13) | 8 (8) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 62 (100) | 53 (76) | 4 (4) | 7 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 12 (12) | 0 (0) | 2 (2)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4) | 2 (2) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 38 (43) | 22 (32) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 31 (32) | 28 (32) | 0 (0) | 2 (2)
Peripheral venous disease (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Patients in this study had to complete treatment in predecessor studies. Therefore selection bias may exist. Baseline is defined for this study's entry value, not all values are prior to active treatment due to some patients being treated previously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT02258542/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT02258542/SAP_001.pdf